CLINICAL TRIAL: NCT04804787
Title: Emotions Recognition in Multiple Sclerosis
Brief Title: Emotions in Multiple Sclerosis
Acronym: RECODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P00107
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Emotions recognition; Cognitive disorders
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: 1 experimental group composed of patients with multiple sclerosis
  1 control group composed of volunteers matched in gender, age, and education's level with the experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group : patients with multiple sclerosis (Experimental): The experimental group will be constituted of patients with multiple sclerosis.
  Interventions: Diagnostic Test: Carrying out a tests and questionnaires battery
- Control group : volunteers (Active Comparator): The control group will be constituted of healthy volunteers with the same characteristics concerning age, sex, education's level as experimental group's patients
  Interventions: Diagnostic Test: Carrying out a tests and questionnaires battery

INTERVENTIONS:
Diagnostic Test: Carrying out a tests and questionnaires battery — The attendees will carry out different questionnaires and tests to evaluate their potential cognitive disorders

SUMMARY:
Through this study, a group composed of multiple sclerosis patients will be compared to a healthy volunteers group to determine if the positive emotions recognitions is preserved in the first group.

DETAILED DESCRIPTION:
Different studies have highlighted the specific deficiency concerning emotions recognition in multiple sclerosis. Patients with multiple sclerosis are reported to have more difficulty recognising negative emotions, especially anger and fear.

In this context, RECODE study has a twofold objective:

* To determine whether the positive emotions recognition remains preserved by combining behavioural and neurophysiological measures (electrodermal activity).
* To study this disorder's etiology through a comparison between a multiple sclerosis patient group and a control group (matched in sex, age, and education's level).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years old.
* Understand and able to express themselves in French.
* EXPERIMENTAL GROUP :
* Relapsing-remitting form (RRMS)
* With an EDSS < 4 (Expanded Disability Status Scale)
* No significant motor, cerebellar or somatosensory disorders of the upper limbs or visual disorders (EDSS specific parameter <2)
* No flare-up in the last 6 weeks
* No corticosteroids taken in the last 4 weeks
* CONTROL GROUP :
* Lack of global cognitive deterioration (according to Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) standards).
* Gender, age and education level matching to the multiple sclerosis patients
* Understanding and signing the informed consent and information letter regarding participation in the study.
* Benefiting from health insurance coverage.

Exclusion Criteria:

* Persons with previous neurological pathologies, head trauma with loss of consciousness, psychiatric pathologies, serious general affections, perceptive or dysarthric disorders preventing verbal communication or reading,
* People with sensory disorders (visual and auditory) that interfere with the performance of neuropsychological tests;
* Treatment with psychotropic drugs (except benzodiazepines and hypnotics).
* Refusal to participate after clear and fair information about the study.
* Major persons under guardianship, under judicial protection, persons deprived of liberty.
* Pregnant or breastfeeding women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Emotion's valence | Day 0
  Through the emotion recognition test, the attendees will have to evaluate the emotion's valence conveyed by the stimuli on a scale ranging from 1 (the emotion conveyed is negative) to 10 (the emotion conveyed is positive).
Emotion's intensity | Day 0
  Through the emotion recognition test, the attendees will have to evaluate the emotion's intensity conveyed by the stimuli on a scale ranging from 1 (the emotion conveyed is not very intense) to 10 (the emotion conveyed is very intense).
Emotion recognition | Day 0
  Comparison of the answers obtained to the recognition question "In your opinion what is the emotion conveyed by this extract/face" in both groupsThrough the emotion recognition test, the attendees will have to evaluate the emotion perceived among 6 basic emotions (anger, disgust, joy, fear, surprise, sadness) and 14 complex emotions (benevolence, disappointment, boredom, enthusiasm, mischief, pride, frustration, shame, hostility, worry, interest, jealousy, sorrow, sneakiness).
Certainty's degree of answers | Day 0
  Certainty's degree of the attendees answers to the recognition question on a scale from 1 ("I am not at all certain of my answer") to 10 ("I am quite certain of my answer")

SECONDARY OUTCOMES:
California Verbal Learning Test (CVLT) | Day 0
  Learning test of a 16 words list belonging to 4 distinct semantic categories (flowers, fish, clothes, fruit). The list is presented 5 times to the patient who must remember it immediately after each presentation, after the presentation of a second interfering list and after a 20-minute delay. A main score is extracted determining how many errors are made in each learning task.
Brief Visuo-spatial Memory Test (BVMT) | Day 0
  Learning test in episodic visuo-spatial memory of 6 simple geometrical drawings. This test presents 3 presentation phases during which the sheet containing the 6 drawings is presented to the participant for 10 seconds, followed by an immediate recall phase (free hand reproduction of the drawings). A delayed recall phase (at 7 minutes) and a delayed recognition phase (among 12 distractors) is also proposed. A main score is extracted.
Symbol Digit Modalities Test (SDMT) | Day 0
  Coding test in which the patient has 90 seconds to state orally the correspondence of numbers (from 1 to 9) to 9 different symbols (matched according to a matching standard). The correct answers number is measured.
Stroop test | Day 0
  The Stroop test is used to evaluate executive functions, especially inhibition abilities and sensitivity to interference. This test offers 3 situations in which performance is measured by the time taken by the patient for each situation and the number of uncorrected errors.
Trail Making test | Day 0
  The Trail Making Test is used to evaluate executive functions especially the cognitive flexibility abilities. The subject's performance is evaluated by the time taken by the subject, the total number of errors and the number of perseveration errors.
Verbal fluency test | Dat 0
  The verbal fluency test evaluates executive functions, and more specifically the spontaneous flexibility's abilities. The performance is evaluated by the number of different words cited.
Beck Depression Inventory (BDI) | At the unique experimental session
  The Beck Depression Inventory is used to assess depressive disorders. It is a 13-items self-questionnaire rated from 0 (no problem) to 3 (maximum severity of this symptom). The depression's severity is assessed by classifying the total score into 3 levels of intensity: <3: Normal; 3-8: Borderline; >8: Depressed.
State Trait Anxiety Inventory Y-A (STAI Y-A) | Day 0
  The STAI Y-A anxiety scale (state anxiety) is used to assess the attendees state anxiety's level. The anxiety's severity is measured by 5 intensity's levels : 35: Very low anxiety; 36-45: Low anxiety; 46-55: Moderate anxiety; 56-65: High anxiety; > 65: Very high anxiety.
State Trait Anxiety Inventory Y-B (STAI Y-B) | Day 0
  The STAI Y-B anxiety scale (trait anxiety) is used to assess the attendees trait anxiety's level. The anxiety's severity is measured by 5 intensity's levels : 35: Very low anxiety; 36-45: Low anxiety; 46-55: Moderate anxiety; 56-65: High anxiety; > 65: Very high anxiety.
Toronto Alexithymia Scale-20 (TAS-20) | Day 0
  The TAS-20 is used to assess the attendees alexithymia's level. The alexithymic syndrome's severity is measured in 4 intensity's levels based on responses to 20 items: 0-51: no alexithymia; 52-60: mild alexithymia; > 60: severe alexithymia.
Dot Probe Task | Day 0
  Through the Dot Probe Task, it is possible to find out whether participants tend to focus their attention on positive or negative information. The reaction time to complete the task and the accuracy of the response are measured.
Change in the electrodermal response during emotion recognition test | Day 0
  Before the emotion recognition test a first resting measurement of the electrodermal response is performed. Then, the attendee electrodermal response will be recorded during the test for each emotional stimulus. At the end of the test, a second resting measurement of the electrodermal response will be performed. The signals obtained during the task will be compared with the attendee resting signals.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Lenne, Principal Investigator — Hôpital Saint Vincent de Paul, Lille
Locations (1):
- Hôpital Saint-Vincent de Paul, Lille, France

IPD SHARING:
Plan to Share IPD: No